CLINICAL TRIAL: NCT04178187
Title: The Role of Probiotics in the Eradication of Helicobacter Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Consultant Gastroenterology, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 444/23/07/2019
Record Dates: First submitted 2019-11-08; First posted 2019-11-26 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; Probiotics; Eradication treatment of H.Pylori; Antibiotics; Proton pump inhibitors; Saccharomyces boulardii; Bifidobacterium lactis; Lactobacillus acidophilus; Lactobacillus plantarum
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactolevure (Active Comparator): Patients will receive quadruple eradication therapy for Helicobacter Pylori infection with Amoxicillin, Clarithromycin, Metronidazole, Omeprazole and Probiotics
  Interventions: Drug: Caps Lactolevure
- Placebo (Placebo Comparator): Patients will receive quadruple eradication therapy for Helicobacter Pylori infection with Amoxicillin, Clarithromycin, Metronidazole, Omeprazole and Placebo
  Interventions: Drug: Caps Placebo

INTERVENTIONS:
Drug: Caps Lactolevure — One group will receive Caps Lactolevure x2 and the other group Caps Placebo x2.
  Other Names: Probiotics
  Arms: Lactolevure
Drug: Caps Placebo — Caps Placebo
  Arms: Placebo

SUMMARY:
All patients will receive quadruple eradication therapy for 10 days with Omerazole 20mg x2, Amoxicilin 1g x2, Clarithromycin 500mg x2 and Metronidazole 500mg x2. The patients will be randomised into two groups. The first group will receive one capsule of probiotics x2 two hours before or after meal for 15 days and the second group placebo (capsule with same composition and colour with probiotic) x2, two hours before or after meal for 15 days as well.

The probiotic (Lactolevure, Uni-Pharma, Athens) contains four probiotic strains known for their effectivness and safety, Saccharomyces Boulandrii (1.5 BU/capsule), Bifidobacterium Lactis BB-12 (1.75 BU/capsule), Lactobacillus Acidodophilus LA-5 (1.75 BU/capsule) and Lactobacillus Plantarum (0.5 BU/capsule).

DETAILED DESCRIPTION:
Patients with H.Pylori infection establised after a uper GI endoscopy and gastric biopsy will receive quadruple eradication therapy for 10 days with Omerazole 20mg x2, Amoxicilin 1g x2, Clarithromycin 500mg x2 and Metronidazole 500mg x2. The patients will be randomised into two groups. The first group will receive one capsule of probiotics x2 two hours before or after meal for 15 days and the second group placebo (capsule with same composition and colour with probiotic) x2, two hours before or after meal for 15 days as well.

The probiotic contains four probiotic strains known for their effectivness and safety, Saccharomyces Boulandrii (1.5 BU/capsule), Bifidobacterium Lactis BB-12 (1.75 BU/capsule), Lactobacillus Acidodophilus LA-5 (1.75 BU/capsule) and Lactobacillus Plantarum (0.5 BU/capsule).

Patients will report in a specific questionnare the presence or absence of symptoms suggestive of side effects associated with the Abx administered (i.e flatulance, abdominal pain, diarrhoea, regurgitation, vomiting).

All patints will be subjected to urea breath test one month after the completion of treatment in order to verify HP eradication.

ELIGIBILITY:
Inclusion Criteria:

* Established Helicobacter Pylori Infection

Exclusion Criteria:

* Pregnancy
* Lactate
* Previous eradication therapy for HP.
* Course of antibiotics and/or probiotics one month prior to stydy entry
* Course of PPI's, H2- antagonst and antacids two weeks prior to study entry
* Known allergy to antibiotics that will be used in study
* Coronary disease, heart failure,malignancy,thyroid disease, pulmonary disease or other serious disease as per medical judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Prevention of antibiotic side effects | Through study completion, an average of 1 year
  Primary prevention of Abx side effects as assessed by a questionnaire including all possible side effects (i.e. vomiting, diarrhea, flatulence etc) on a ten point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Viazis, Dr, Principal Investigator — Evangelismos Hospital; Katerina Kotzampassi, MD, Principal Investigator — AHEPA University Hospital; Olga Giouleme, MD, Principal Investigator — General Hospital Of Thessaloniki Ippokratio; Periklis Apostolopoulos, MD, Principal Investigator — NIMTS Hospital; Sotirios Georgopoulos, MD, Principal Investigator — Iatriko Palaiou Falirou
Locations (5):
- Greece (5):
  - Evangelismos Hospital, Athens, Attica
  - NIMTS Hospital, Athens
  - Iatriko Palaiou Falirou, Palaió Fáliro
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
  - General Hospital of Thessaloniki Ippokratio, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kotzampassi K, Stavrou G, Damoraki G, Georgitsi M, Basdanis G, Tsaousi G, Giamarellos-Bourboulis EJ. A Four-Probiotics Regimen Reduces Postoperative Complications After Colorectal Surgery: A Randomized, Double-Blind, Placebo-Controlled Study. World J Surg. 2015 Nov;39(11):2776-83. doi: 10.1007/s00268-015-3071-z. PMID 25894405